CLINICAL TRIAL: NCT02172768
Title: Pharmacokinetics of Micafungin (Mycamin ®) as Antifungal Prophylaxis Given Twice Weekly Intravenously Compared to Micafungin Given Daily to Patients at Risk for Developing an Invasive Fungal Disease.
Brief Title: Pharmacokinetics of Micafungin Given Twice Weekly Intravenously Compared to Micafungin Given Daily to Patients at Risk for Developing an Invasive Fungal Disease
Acronym: MATADOR
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: MATADOR
Record Dates: First submitted 2014-06-20; First posted 2014-06-24 (Estimated); Last update posted 2020-12-08 (Actual); Status verified 2020-12

CONDITIONS: Acute Graft Versus Host Disease Grade II-IV; Allogeneic Stem Cell Transplant; Acute Myeloid Leucaemia; Myelo Dysplastic Syndrome
Keywords: pharmacokinetics; alternate dosing; micafungin
MeSH Terms: interventions — Micafungin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- alternate dosing (Experimental): treatment for 8 days with intravenous micafungin twice weekly
  Interventions: Other: alternate dosing; Drug: micafungin
- daily dosing (Active Comparator): micafungin daily for 8 days
  Interventions: Other: daily dosing; Drug: micafungin

INTERVENTIONS:
Other: alternate dosing — treatment for 8 days with intravenous micafungin twice weekly
  Other Names: micafungin
  Arms: alternate dosing
Other: daily dosing — micafungin daily for 8 days
  Arms: daily dosing
Drug: micafungin

SUMMARY:
The primary objective of this trial is as follows:

To determine the pharmacokinetics of micafungin given twice weekly in patients at risk for developing an invasive fungal disease (patients who are being treated for acute or chronic graft versus host disease; patients receiving reduced intensity conditioning for Stem Cell Transplant (SCT); receiving first remission induction chemotherapy for Acute Myeloid Leucaemia (AML)/MyeloDysplasticSyndrome (MDS)) compared to the pharmacokinetics of micafungin given daily.

The secondary objective of this trial is as follows:

To determine whether adequate exposure of micafungin is attained. To determine the safety of micafungin in this patient population

DETAILED DESCRIPTION:
Micafungin has been shown to be a reasonable option for treating invasive aspergillosis in hematopoietic stem cell transplantation (HSCT) recipients and has proven as effective as fluconazole for prophylaxis. Whilst micafungin has much to offer, little is known about its pharmacokinetic profile in specific patient populations, specifically concerning alternate dosing strategies with increased dosages over a prolonged dosing interval. Sufficient data are lacking up to now for twice weekly administration of micafungin as antifungal prophylaxis. Decreasing the dosing frequency to twice weekly seems a reasonable approach considering the long terminal elimination life (i.e. 10-17 h) and considering the data available from murine models that support the use of less frequent dosing with higher dosages.

It will enable us to characterize both the pharmacokinetics of micafungin in the hematology cohort and directly compare the exposure to the alternate dosing strategy.

ELIGIBILITY:
Inclusion Criteria:

* Patient receives immunosuppressive therapy for acute GvHD grade II-IV or reduced intensity conditioning regimens for allogeneic stem cell transplant, or patients receiving first remission induction chemotherapy for AML/MDS.
* Subject is at least 18 of age on the day of providing informed consent.
* Has no signs or symptoms of invasive fungal disease
* If a woman, is neither pregnant nor able to become pregnant and is not nursing an infant.
* Less than 1 week of immunosuppressive therapy for grade II-IV acute GvHD.
* Is managed with a central venous catheter (preferably a quadruple Arrow-Howes™ Quad-Lumen 8.5,5 French; Arrow International).
* Subject is able and willing to sign the Informed Consent before screening evaluations.

Exclusion Criteria:

* Documented history of sensitivity to medicinal products or excipients similar to those found in the micafungin preparation.
* History of or current abuse of drugs, alcohol or solvents.
* Inability to understand the nature of the trial and the procedures required.
* Has not previously participated in this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-10; Primary Completion 2016-06 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
area under the curve | day 4 and day 8
  Full pharmacokinetic curves will be taken op Day 4 or 5 and Day 8 (micafungin). AUC of two dosing regimens will be compared.

SECONDARY OUTCOMES:
population PK model | Day 4 and Day 8
  to perform Monte Carlo simulations to provide the scientific background for alternate dosing strategies in the prophylactic setting
adverse events | day 1- 11
  number and severity of adverse events will be recorded during the study and both treatment regimens will be compared

CONTACTS AND LOCATIONS:
Overall Officials: Roger Brüggemann, Principal Investigator — Radboud University Medical Center
Locations (2):
- UZ Leuven, Leuven, Belgium
- Radboudumc, Nijmegen, Netherlands

REFERENCES:
- [Result] Muilwijk EW, Maertens JA, van der Velden WJFM, Ter Heine R, Colbers A, Burger DM, Andes D, Theunissen K, Blijlevens NMA, Bruggemann RJM. Pharmacokinetics of extended dose intervals of micafungin in haematology patients: optimizing antifungal prophylaxis. J Antimicrob Chemother. 2018 Nov 1;73(11):3095-3101. doi: 10.1093/jac/dky324. PMID 30137340